CLINICAL TRIAL: NCT03255096
Title: Open-Label, Dose Escalation/Expansion Phase Ib Study to Evaluate the Safety, Pharmacokinetics, and Clinical Activity of the Combination of RO6870810 and Venetoclax, With or Without Rituximab, in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL) and/or High-Grade B-Cell Lymphoma With MYC and/or BCL2 and/or BCL6 Gene Rearrangements
Brief Title: A Study to Evaluate Safety, Pharmacokinetics, and Clinical Activity of Combination of RO6870810 and Venetoclax, With or Without Rituximab, in Participants With Relapsed/Refractory DLBCL and/or High-Grade B-Cell Lymphoma and/or High Grade B-Cell Lymphoma With MYC and/or BCL2 and/or BCL6
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP39461; 2017-000357-39 (EudraCT Number)
Record Dates: First submitted 2017-07-31; First posted 2017-08-21 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Diffuse Large B-cell Lymphoma; High-Grade B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — RO6870810; venetoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Phase (Part 1) (Experimental): Participants will receive either RO6870810 and venetoclax or RO6870810 and venetoclax along with rituximab until disease progression, unacceptable toxicities or withdrawal from treatment for other reasons, or death.
  Interventions: Drug: RO6870810; Drug: Venetoclax; Drug: Rituximab
- Expansion Phase (Part 2) (Experimental): Participants will receive RO6870810 and venetoclax along with rituximab (or RO6870810 and venetoclax, if the combination of the 3 drugs is not tolerable) at a recommended dose established in dose escalation phase until disease progression, unacceptable toxicities or withdrawal from treatment for other reasons, or death.
  Interventions: Drug: RO6870810; Drug: Venetoclax; Drug: Rituximab

INTERVENTIONS:
Drug: RO6870810 — RO6870810 subcutaneously (SC) at dose of 0.30, 0.45, or 0.65 milligram per kilogram (mg/kg) on Days 1-14 of 21-day cycles.
Drug: Venetoclax — Venetoclax tablets orally at dose of 400 mg once daily (QD) continuously for 21 days.
Drug: Rituximab — Rituximab intravenously (IV) at dose of 375 mg/m^2 weekly during the first 21-day cycle (C1) and on day 1 of each cycle thereafter.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and clinical activity of RO6870810 in combination with venetoclax and when co-administered with rituximab in participants with relapse/refractory (R/R) diffuse large B-cell lymphoma (DLBCL) and/or high-grade B-cell lymphoma with myelocytomatosis oncogene (MYC) and/or B-cell lymphoma 2 (BCL2) and/or B-cell lymphoma 6 (BCL6) gene rearrangements (HGBL-DH/TH).

ELIGIBILITY:
Inclusion Criteria

* Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
* Life expectancy >3 months as per investigator's assessment.
* Part 1 and Part 2 Group 1: Participantts with diffuse large B-cell lymphoma (DLBCL) relapsed or refractory to ≥ 1 course of chemotherapy including an anti-CD20 monoclonal antibody, and not eligible for autologous stem cell transplantation (ASCT) (including due to chemorefractory disease). Participants with transformed FL are eligible, provided DLBCL or HGBL-DH/TH histology is biopsy-confirmed prior to study entry and a treatment regimen as described above has been administered. The Sponsor retains the option to limit the number of participants enrolled with transformed FL.

Part 2, Group 2: Patients identified with DE-DLBCL (expression MYC ≥40%, BCL2 > 50%) and or HGBL-DH/TH, relapsed or refractory to >= 1 course of chemotherapy including an anti-CD20 monoclonal antibody, and not eligible for ASCT (including due to chemorefractory disease). Patients with transformed follicular lymphoma (FL) are eligible, provided DE-DLBCL and/or HGBL-DH/TH histology is biopsy-confirmed prior to study entry and a treatment regimen as described above has been administered. The Sponsor retains the option to limit the number of participants enrolled with transformed FL.

* Part 1 and Part 2: Willing to provide the protocol specified tumor biopsy(ies): at screening a fresh biopsy (if no archival biopsy tissue of less than 3 months prior to treatment and without intercurrent treatment is available); Part 2: Willing to provide an additional biopsy on Cycle 2 Day 15 (+ 2 days).
* Acceptable liver function, as specified below:

  * Total bilirubin ≤ 2 times upper limit of normal (ULN). (Participants with known Gilbert's disease who has serum bilirubin ≤ 3 × ULN may be enrolled).
  * Aspartate transaminase (AST; SGOT), alanine transaminase (ALT; SGPT) ≤ 2.5 × ULN, (or ≤ 5 × ULN if tumor involvement (liver) is present).
  * Gamma-glutamyl transferase (GGT) alkaline phosphatase ≤ 2.5 × ULN.
* Acceptable renal function, as specified below:

  • Creatinine clearance (CrCl) calculated by Cockroft-Gault formula of ≥ 60 mL/min.
* Acceptable hematologic status (growth factors cannot be used within the previous 7 days), as specified below:

  * Absolute neutrophil count (ANC) ≥ 1000 cells/μL
  * Hemoglobin ≥ 9 g/dL
  * Platelet count ≥ 75,000 (platelets/μL)
* Uncontrolled symptomatic hypercalcemia.
* Acceptable coagulation status, as specified below:

  * Prothrombin time (PT) and partial thromboplastin time (PTT) ≤ 1.2 × ULN (unless receiving anticoagulation therapy, if receiving anticoagulation therapy, eligibility will be based upon international normalized ratio [INR]).
  * INR ≤ 1.6 (unless receiving anticoagulation therapy).
  * If receiving warfarin: INR ≤ 3.0 and no active bleeding (i.e., no bleeding within 14 days prior to first dose of study therapy).
* Acceptable method of contraception

Exclusion Criteria

* Current central nervous system (CNS) lymphoma or leptomeningeal infiltration.
* New York Heart Association (NYHA) Class III or IV cardiac disease, myocardial infarction, within the past 6 months, unstable arrhythmia, or known pericardial disease.
* Fredericia-corrected QT interval (QTcF) >470 msec (female) or >450 msec (male), or history of congenital long QT syndrome.
* Any electrocardiogram (ECG) abnormality, which in the opinion of the Investigator would preclude safe participation in the study.
* Active, uncontrolled bacterial, viral, or fungal infections, within 7 days of study entry requiring systemic therapy.
* Clinically important respiratory impairment
* Grade ≥ 3 sensory or motor neuropathy.
* Any Grade >1 (according to the NCI CTCAE 4.03) adverse reaction unresolved from previous treatments and not readily managed and controlled with supportive care.
* Serious non-malignant disease that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.
* History of progressive multifocal leukoencephalopathy (PML).
* History of other malignancy within 2 years prior to screening, except for ductal carcinoma in situ not requiring chemotherapy, appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, low-grade, localized prostate cancer (Gleason score ≤ 7) not requiring treatment or appropriately treated Stage I uterine cancer.
* Completion of ASCT within 100 days prior to Day 1 of Cycle1.
* Prior standard or investigational anti-cancer therapy, as specified below:

  * Radio-immunoconjugate 4 weeks or 5 half-lives, whichever is longer prior to Day 1 of Cycle 1.
  * Monoclonal antibody or antibody-drug conjugate (ADC) therapy within 3 weeks prior to Day 1 of Cycle 1.
  * Radiotherapy, chemotherapy, or targeted small-molecule therapy within 2 weeks prior to Day 1 of Cycle 1.
  * CAR T-cell therapy 30 days prior to Day 1 of Cycle 1.
* History of major solid organ transplant (i.e., heart, lungs, liver and kidney).
* History of an allogeneic bone marrow transplant.
* Major surgical procedure within 28 days prior to Day 1 of Cycle 1.
* Treatment with systemic corticosteroids ≥ 20 mg/day prednisone or equivalent, for non-lymphoma treatment reasons. For lower acceptable doses, documentation of a stable dose for at least 4 weeks prior to Day 1 of Cycle 1 is required.

  18. Treatment with strong to moderate CYP3A inhibitors or moderate CYP3A inducers within 7 days prior to the first dose of study treatment.
* Treatment with strong CYP3A inducers within 14 days prior to the first dose of study treatment of RO6870810/venetoclax.
* Consumption of grapefruits, grapefruit products, Seville oranges (including marmalade that contains Seville oranges), or star fruit within 3 days prior to the first dose of venetoclax.
* Participants who are currently receiving any other investigational agent ((other than anti-cancer therapy as specified in exclusion criteria number 13) or have received an investigational agent within 30 days or 5 half-lives prior to Day 1 of Cycle 1, whichever is longer.
* Prior treatment with small molecule bromodomain and extra terminal (BET) family inhibitor.
* Known to be human immunodeficiency virus (HIV) positive.
* Presence of positive test results for hepatitis B surface antigen (HBsAg) or hepatitis C antibodies (HcAb) (for participants receiving regimen including rituximab)
* Pregnant or breastfeeding female.
* Significant allergy to a biological pharmaceutical therapy that, in the opinion of the Investigator, poses an increased risk to the participant.
* Uncontrolled cancer pain. Participants requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions amenable to palliative radiotherapy should be treated prior to enrollment.
* History of severe allergic or anaphylactic reaction to humanized or murine monoclonal antibodies (for participants receiving regimen including rituximab).
* Known sensitivity or allergy to murine products or any component of RO6870810, venetoclax, or rituximab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose-Limiting Toxiciities (DLT)- Part 1 | Cycle (C) 1 (21 days)
  DLT is defined as any of the toxicities- occurs within the first cycle for which the participant receives the full intended combination doses and number of administrations; is considered to be related to study treatment by the investigator; is not attributed to disease progression or another clearly identifiable cause.
Percentage of Participants With Adverse Events (AEs) - Part 1 | Up to 36 months
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Percentage of Participants With Clinically Significant Changes in Vital Signs, Physical Examination, Clinical Laboratory Results and Electrocardiogram (ECG) Findings- Part 1 | Up to 36 months
Complete Response (CR) Rate as Determined by Independent Radiological Central Review (ICR) Using Modified Lugano Response Criteria- Recommended Dose (RD) Expansion - Part 2 | Up to 36 months
Overall Response (OR) Rate as Determined by Independent Radiological Central Review (ICR) Using Modified Lugano Response Criteria- RD Expansion - Part 2 | Up to 36 months

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) - Part 2 | Up to 36 months
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Percentage of Participants With Clinically Significant Changes in Vital Signs, Physical Examination, Clinical Laboratory Results and Electrocardiogram (ECG) Findings- Part 2 | Up to 36 months
Maximum Concentration (Cmax) of RO6870810 and its Potential Metabolites- Part 1 and Part 2 | Pre-dose Day 1,8,15; 0.25,0.5,1,2,4,6,8 hour (h) post-dose Day 1, 15; Day 2 C1; Pre-dose Day 1,8,15; 0.25h post-dose Day 1,8 C2; Pre-dose Day 1,15 C4; 0.25h post-dose Day 1 C4; Pre-dose, 0.25h post-dose Day 1 of subsequent even Cycles (Up to 36 months)
Trough Serum Concentration (Cmin) of RO6870810 and its Potential Metabolites- Part 1 and Part 2 | Pre-dose Cycle 2 and all other subsequent even Cycles (Up to 36 months)
Time of Maximum Concentration (tmax) of RO6870810 and its Potential Metabolites- Part 1 and Part 2 | Pre-dose Day 1,8,15; 0.25,0.5,1,2,4,6,8 hour (h) post-dose Day 1, 15; Day 2 C1; Pre-dose Day 1,8,15; 0.25h post-dose Day 1,8 C2; Pre-dose Day 1,15 C4; 0.25h post-dose Day 1 C4; Pre-dose, 0.25h post-dose Day 1 of subsequent even Cycles (Up to 36 months)
Clearance (CL) of RO6870810 and its Potential Metabolites- Part 1 and Part 2 | Pre-dose Day 1,8,15; 0.25,0.5,1,2,4,6,8 hour (h) post-dose Day 1, 15; Day 2 C1; Pre-dose Day 1,8,15; 0.25h post-dose Day 1,8 C2; Pre-dose Day 1,15 C4; 0.25h post-dose Day 1 C4; Pre-dose, 0.25h post-dose Day 1 of subsequent even Cycles (Up to 36 months)
Volume of Distribution (Vd) of RO6870810 and its Potential Metabolites- Part 1 and Part 2 | Pre-dose Day 1,8,15; 0.25,0.5,1,2,4,6,8 hour (h) post-dose Day 1, 15; Day 2 C1; Pre-dose Day 1,8,15; 0.25h post-dose Day 1,8 C2; Pre-dose Day 1,15 C4; 0.25h post-dose Day 1 C4; Pre-dose, 0.25h post-dose Day 1 of subsequent even Cycles (Up to 36 months)
Area Under the Curve (AUC) of RO6870810 and its Potential Metabolites- Part 1 and Part 2 | Pre-dose Day 1,8,15; 0.25,0.5,1,2,4,6,8 hour (h) post-dose Day 1, 15; Day 2 C1; Pre-dose Day 1,8,15; 0.25h post-dose Day 1,8 C2; Pre-dose Day 1,15 C4; 0.25h post-dose Day 1 C4; Pre-dose, 0.25h post-dose Day 1 of subsequent even Cycles (Up to 36 months)
Complete Response (CR) Rate as Determined by the Investigator Based on the Modified Lugano Response Criteria- Part 1 and Part 2 | Up to 36 months
Complete Response (CR) Rate, as Determined by the ICR and by the Investigator on the Basis of CT Scans Alone- Part 1 and Part 2 | Up to 36 months
Objective Response Rate, as Determined by the ICR and by the Investigator on the Basis of Modified Lugano Response Criteria- Part 1 and Part 2 | Up to 36 months
Objective Response Rate, as Determined by the ICR and by the Investigator on the Basis of CT Scans Alone- Part 1 and Part 2 | Up to 36 months
Duration of Response (DoR)- Part 1 and Part 2 | Up to 36 months
Progression-Free Survival (PFS)- Part 1 and Part 2 | Up to 36 months
Event-Free Survival (EFS)- Part 1 and Part 2 | Up to 36 months
Disease-Free Survival (DFS)- Part 1 and Part 2 | Up to 36 months
Overall Survival (OS)- Part 1 and Part 2 | Up to 36 months
Half-Life (t1/2) of RO6870810 and its Potential Metabolites- Part 1 and Part 2 | Pre-dose Day 1,8,15; 0.25,0.5,1,2,4,6,8 hour (h) post-dose Day 1, 15; Day 2 C1; Pre-dose Day 1,8,15; 0.25h post-dose Day 1,8 C2; Pre-dose Day 1,15 C4; 0.25h post-dose Day 1 C4; Pre-dose, 0.25h post-dose Day 1 of subsequent even Cycles (Up to 36 months)
Percentage of Ant-Drug Antibodies (ADA) Against Rituximab - Part 1 and Part 2 | Pre-dose, End of Infusion Day 1 Cycle 1; Pre-dose Day 1 Cycle 2, 3, 4 , 6 and all other even Cycles (Up to 36 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (9):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - Weill Cornell Medical College, New York, New York
  - Levine Cancer Institute - Blythe, Charlotte, North Carolina
- Peter MacCallum Cancer Centre-East Melbourne, Melbourne, Victoria, Australia
- Rigshospitalet; Hæmatologisk Klinik, København Ø, Denmark
- Spain (3):
  - Hospital de la Santa Creu i Sant Pau; Servicio de Hematologia, Barcelona
  - Hospital Duran i Reynals; Servicio de Hematologia, Barcelona
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid

REFERENCES:
- [Derived] Dickinson M, Briones J, Herrera AF, Gonzalez-Barca E, Ghosh N, Cordoba R, Rutherford SC, Bournazou E, Labriola-Tompkins E, Franjkovic I, Chesne E, Brouwer-Visser J, Lechner K, Brennan B, Nuesch E, DeMario M, Ruttinger D, Kornacker M, Hutchings M. Phase 1b study of the BET protein inhibitor RO6870810 with venetoclax and rituximab in patients with diffuse large B-cell lymphoma. Blood Adv. 2021 Nov 23;5(22):4762-4770. doi: 10.1182/bloodadvances.2021004619. PMID 34581757